CLINICAL TRIAL: NCT03204591
Title: Risk of Bacterial Infection in Cirrhotic Patients With Acute Severe Liver Injury: a Multicenter,Prospective, Observational Study
Brief Title: Bacterial Infections in Cirrhotic Patients With Acute Severe Liver Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Zhejiang Study Group for Organ Failure in Cirrhosis (Other)
Collaborators: Ningbo No.2 Hospital (Other)
Responsible Party: Principal Investigator, Shi Yu, Principal Investigator, The Zhejiang Study Group for Organ Failure in Cirrhosis
Other Study IDs: NSFC81670567
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Cirrhosis, Liver; Bacterial Infections; Acute Liver Injury
MeSH Terms: conditions — Liver Cirrhosis; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LC with SALI: cirrhosis patients with severe acute liver injury
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Acute hepatic insults including hepatitis flare-up, active alcohol assumption and hepatotoxic drug use are common in patients with cirrhosis especially in Eastern countries.These patients are at high risk of developing acute-on-chronic liver failure (ACLF) and associated with high short-term mortality. And the natural history of these patients is frequently complicated by bacterial infections, which lead to deterioration of underlying diseases. The present study is aimed to investigate the prevalance and risk factors of bacterial infections in those patients and its impact on in-hospital/short-term mortality.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of cirrhosis confirmed by liver biopsy, endoscopy, radiological examination, or clinical evidence of prior hepatic de-compensation;
2. Flare up of acute severe liver injury within one month before enrollment. Acute severe liver injury is defined as: increase of serum bilirubin >=85mmol/L and international normalized ratio (INR)>=1.5 with a definite hepatic insult.

Exclusion Criteria:

(1)pregnancy; (2) disseminated maliganancy; (3)previously received a liver transplant; (4) HIV infection;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cirrhosis of any etiology who had acute severe liver injury
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-10-18 (Estimated); Study Completion 2019-01-18 (Estimated)

PRIMARY OUTCOMES:
Occurrence of bacterial infection | Within 3 months from admission
  Site,source, pathogen and severity

SECONDARY OUTCOMES:
28-day Mortality | Within 28 days after enrollment
  Disease-associated mortality
90-day Mortality | Within 90 days after enrollment
  Disease-associated mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jifang Sheng, Doctor, Study Chair — Department of infectious disease, First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No